CLINICAL TRIAL: NCT06883292
Title: The Effects of Tyrosol and Creatine on Endurance, Strength, and Fatigue Resistance in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Effects of Tyrosol and Creatine on Endurance, Strength, and Fatigue Resistance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00084231
Record Dates: First submitted 2025-02-27; First posted 2025-03-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Tyrosol; Creatine; Endurance Performance; Cognition
Keywords: tyrosol; creatine; muscle strength; muscle endurance; muscle recovery; muscle performance; reaction time
MeSH Terms: interventions — 4-hydroxyphenylethanol; Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tyrosol and Creatine (Experimental): creatine and tyrosol (3g creatine monohydrate + 500mg tyrosol/day) administered daily
  Interventions: Dietary Supplement: Tyrosol; Dietary Supplement: Creatine
- Tyrosol + placebo (Experimental): 500mg Tyrosol (administered daily as 1 capsule, containing 500mg/capsule) + 3g of resistant dextrin powder (placebo)
  Interventions: Dietary Supplement: Tyrosol; Dietary Supplement: Resistant Dextrin
- Creatine + placebo (Active Comparator): 3g Creatine Monohydrate powder + 500mg Resistant dextrin capsules (as 1 capsule, containing 500mg/capsule) (placebo) administered daily
  Interventions: Dietary Supplement: Creatine; Dietary Supplement: Resistant Dextrin
- placebo + placebo (Placebo Comparator): 3g of resistant dextrin powder (placebo) + 500mg Resistant dextrin capsules (administered as 1 capsule, containing 500mg/capsule) (placebo) administered daily
  Interventions: Dietary Supplement: Resistant Dextrin

INTERVENTIONS:
Dietary Supplement: Tyrosol — phenolic compound found in olive oil
  Arms: Tyrosol + placebo; Tyrosol and Creatine
Dietary Supplement: Creatine — chemical produced naturally by the body used to rapidly regenerate ATP
  Arms: Creatine + placebo; Tyrosol and Creatine
Dietary Supplement: Resistant Dextrin — A type of soluble dietary fiber that is resistant to digestion in the small intestine. It is a byproduct of the starch hydrolysis process, where starch is broken down into smaller chains of glucose molecules
  Arms: Creatine + placebo; Tyrosol + placebo; placebo + placebo

SUMMARY:
The purpose of this clinical trial is to look at tyrosol's effects on endurance, strength, and fatigue resistance in humans. Additionally, the combination of tyrosol and creatine monohydrate will also be looked at to determine if there is a cooperative effect from using both together. It will be conducted over a 4-week period to compare the effects of the following substances: 1) tyrosol, 2) a placebo (a look-alike substance that contains no drug), 3) creatine, and 4) a combination containing both creatine and tyrosol. Endurance, strength, and fatigue resistance will be compared between groups through repeated testing (described below).

Participants who pass initial screening will be invited on-site for day one (Visit 1) of testing where they will proceed with a series of tests which will include the following: (1) body composition; (2) cognitive testing; (3) full-body strength testing; (4) grip strength on both hands; (5) muscle power testing; (6 & 7) Resting blood lactic acid testing followed by 5RM (repetition maximum) bench press, leading to multiple sets of bench press (based on the previous weight) completed to failure, followed by another blood lactic acid reading; (8) a repeat of the muscle power testing; (9) a 1 mile time trial run completed as fast as possible.

After the 4-week supplementation period (~28-34 days), all original measures will be repeated as before in the same order (Visit 2). Approximately 24 hours later (Visit 3) participants will then repeat all physical testing procedures except tests 1, 6, 7, and 8, to determine physical recovery. Additionally, questionnaires for soreness and perceived recovery will also be completed at the beginning of Visit 2 and 3, and again on its own as the only testing event at 48 hours post-Visit 2 (visit 4).

DETAILED DESCRIPTION:
This study will be a randomized, double-blind, placebo-controlled trial. It will be conducted over a 4-week intervention investigating the effects of tyrosol (500mg Tyrosol); placebo control (3g resistant dextrin), and two additional groups including creatine alone (3g creatine monohydrate) and a combination group containing both creatine and tyrosol (3g creatine monohydrate + 500mg tyrosol/day). Endurance, strength, and fatigue resistance will be examined through repeated strength and endurance testing as described below.

On day one (Visit 1) of testing, after a minimum 8-hour overnight fast, subjects will proceed with a series of tests in the following successive order: (1) DXA for body composition followed by consumption of a standardized food bar snack and at least a 15-minute break after the snack. After the 15-minute break, subjects will proceed with the following tests: (2) Psychomotor Vigilance Test (PVT); (3) full-body strength measurement using a computerized mid-thigh pull; (4) strength via grip strength on both hands, tested in triplicate using a dynamometer; (5) 2 sets of 2 plyometric push-ups (with the average of each set used as the outcome metric) on a dual ground-reaction force plate, with a 30 seconds rest between sets; (6 & 7) Resting blood lactate will be measured in duplicate followed by determination of the subject's 5RM (repetition maximum) bench press, which will be used to calculate their 1RM. Subjects will then perform one set of bench at 70% of the calculated 1RM to failure, followed by three sets to failure at 50 % of 1RM with a two-minute rest between all sets. After completion of the last set, another blood lactate reading will be taken (in duplicate) and recorded; (8) subjects will then perform the plyometric push-up protocol one more time to assess the immediate effects of fatigue; (9) subjects will then complete a 1 mile time trial run completed as fast as possible. Rate of Perceived Exertion (RPE) will also be collected during the 1 mile run using Borg RPE scale (Borg, 1982).VO2 max will be estimated from the 1 mile run time, age, gender and BMI, using equations described by Kayihan et al. (2014). Finally, the subjects will repeat the PVT at the end of the session.

After the 4 week supplementation period (approximately 28+6 days), all baseline measures will be repeated in the fasted state, in the same successive order (Visit 2). Approximately 24 hours later (Visit 3) subjects will then repeat all physical testing procedures except tests 1, 6, 7, and 8 (which would exclude DXA, Blood Lactate, Bench Press 5RM and sets to failure, and the second plyometric push-up test) to assess physical recovery between groups. Additionally, likert scales for soreness and perceived recovery will be completed as the first outcome measure just prior to the first PVT exam, at Visit 2 and 3, and again on its own as the only testing event performed at 48 hours post-bout (visit 4). Finally, on post-testing days (Visit 2 and 3), a full dosage of the study treatment will be taken with water, as well as a standardized food bar snack; and will be administered on-site by staff. On visit 2, this supplement will be taken just after completion of the DXA (prior to Likert and PVT); on Visit 3, the treatment will be taken prior to the start of Likert scales and PVT testing. The subjects will wait for at least 15 minutes after the snack and treatment to begin the remaining tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-50
* Currently active (engaged in moderate to vigorous activity at least 2-days per week as defined by the American College of Sports Medicine Guidelines)
* Estimated VO2 max equal to or greater than the 50th percentile of the population norm for age (assessed via ACSM guidelines, 2014). The VO2 max estimation at screening will be obtained by following a non-exercise regression model validated and described by Bradshaw et al. (2005).
* Able to read and write in English
* During the study, agree not to take any other supplements that may increase muscle strength or endurance (e.g. protein formulas, creatine, amino acids, tyrosol or stimulants other than caffeine).
* Females willing to share days menstrual cycle for testing purposes as shifts in hormone levels may, potentially, affect testing

Exclusion Criteria:

* Known diagnosis of any cardiovascular, metabolic, endocrine, or renal disease
* Recent musculoskeletal injury (<3-months)
* Recent orthopaedic surgery (<12-months)
* History or current malignancy
* Previous gastrointestinal surgery within the past 12 months
* Regular smoker
* Regular drinker (>14 drinks per week)
* Current use (within the past 4 weeks) of creatine supplements
* Current use (within past 3 months) of Tyrosol supplementation
* Current use of dietary supplements that may enhance mitochondrial function, muscle hypertrophy, or muscle strength (e.g. protein formulas, creatine, amino acids, tyrosol, etc.).
* Current use of prescription medications that may influence adaptation to exercise (hormone therapies, peptides, etc.)
* Female subjects who do not test negative on a urine pregnancy test or are lactating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Mid Thigh Pull | Performed one time at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3)
  Utilizing a pronated clean grip, subjects will be instructed to assume a body position similar to the second pull of the snatch and clean. Once body positioning is stabilized, the subject will be given a countdown. Minimal pre-tension will be allowed to eliminate slack prior to initiation of the IMTP. Each subject will perform two warm-up reps, one at 50% and one at 75% of perceived maximum effort. Thereafter, subjects will complete two maximal IMTPs separated by approximately two minutes of rest. Force kinematics from the IMTP will be collected and recorded using a linear position transducer.
1-mile run | Performed one time at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3)
  Participants will complete the 1-mile run time trial on a treadmill. The treadmill allows participants to adjust the speed as needed to maintain their maximal sustainable pace throughout the test. The total time taken to complete the 1 mile will be recorded as the primary performance measure.
Rate of Perceived Exertion (RPE) | Performed at 0, 0.25, 0.5, 0.75, and 1.0 miles during the 1-mile run at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3)
  RPE will be collected during the 1 mile run using Borg RPE scale (Borg, 1982). Participants will be asked to select a number on the scale to rate their overall effort. A rating of 6 is said to be no effort (rest) and a rating of 20 is considered to be maximal effort. All perceptual measures will be collected in isolation from other participants to promote accuracy and recorded as arbitrary units (a.u.).
Grip Strength | Performed one time at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3)
  Grip strength will be conducted using a digital hand dynamometer (Vernier Lab). The dynamometer is an isometric force sensor (strain gauge amplifier-based) that measures the force applied to its pressure pads. 5-second maximal voluntary contractions are performed on both of the participant's hands, measured in triplicate. With the subject's back supported and straight, 90 degrees of elbow flexion, and 0 degrees of shoulder flexion, participants hold the dynamometer in the palm and secure a comfortable grip. They are then instructed to squeeze with maximum force which will be measured by the Vernier LabQuest® 2 dynamometer and analyzed using Logger Pro software (Version 3.16.2). Average and peak force values will be utilized for study analysis.
Plyometric Push Up (Force Plate) | Performed 2 times (once before bench press and once after bench press) at baseline (visit 1) and at day 28 (visit 2). AT day 29, this will be performed 1 time (visit 3).
  The force plate is a platform composed of two force plates that separate the platform into left and a right halves. Each plate contains four force sensors which measure the vertical ground reaction force exerted on the platform. The sensors are connected to a laptop computer and analyzed using the Mechanography GRFP Research Edition® software (version 4.2-b05.53-RES).
  For the Plyometric Pushup exercise, subjects will perform two sets of two plyometric push-ups on the force plate. Subjects will assume a push up position with one hand centered on each half of the force plate. Each subject will be given an initiation command by the researcher and then perform two maximal effort plyometric push ups on the force plate, pressing themselves as high as possible into the air on each repetition. Subjects will be given 30sec of rest and then repeat once more. Force curves will be analyzed for peak force, rate of force development, and limb symmetry. Results will be averaged and analyzed.
Bench Press 5 repetition maximum (RM) | Performed one time at baseline (visit 1) and at day 28 (visit 2).
  Subjects will be asked to perform a 5 repetition maximum (RM) lift in order to calculate their 1RM for determination of weight needed for the protocol. They will start with a warm-up consisting of the following: 1 set of 8-10 reps of a light weight of their choosing followed by 1-2 sets of 3-5 reps of progressively heavier weights (~50-70% of self-estimated 1RM). Following a 2-minute rest, subjects will select a weight they feel confident they can do for 5-7 reps but not more than 7 reps (based on warm-up weights). Weight will be increased until the subject is only able to complete 5 reps with good form. This will be their 5RM. For safety, a spotter will always be present for lifts and a set of safety bars will be used as well.
  Subject's 1RM will be calculated from this 5RM using the Brzycki formula (Macarilla CT, et.al. 2022) 1RM = W / (1.0278 - 0.0278 × R), where W represents the weight lifted in pounds, and R represents the number of repetitions.
Bench Press Repetitions to Failure | Performed one time at baseline (visit 1) and at day 28 (visit 2).
  After calculating the estimated 1RM from the 5RM, subjects will then perform one set of bench press at 70% of the calculated 1RM to failure, followed by three sets to failure at 50 % of 1RM with a two-minute rest between all sets. Total repetitions for each of these sets will be recorded and will be used to determine fatigue and compared to follow-up Visit 2 performance for fatigue resistance. For safety, a spotter will always be present for lifts and a set of safety bars will be used as well.

SECONDARY OUTCOMES:
Body Composition (DXA) | Performed one time at baseline (visit 1) and at day 28 (visit 2).
  Total and regional body composition will be determined by a whole-body scan on a dual-energy x-ray absorptiometry device (DXA) (Horizon A DXA System, Hologic Inc, Marlborough, MA). Each subject will be scanned by a certified technician, and the digital segmentation will be determined via computer algorithm. Fat-free mass, fat mass, and body fat percentage will be determined for each scan. Calibration will be performed against a phantom prior to testing. The abdominal region will be delineated by an upper horizontal border located at half of the distance between the acromion processes and external end of iliac crests, a lower border determined by the external end of iliac crests and the lateral borders extending to the edge of the abdominal soft tissue. All trunk tissue within this standardized height region will be selected for analysis.
Blood Lactate | Performed one time at baseline (visit 1) and at day 28 (visit 2).
  Blood lactate will be measured using the Nova Biomedical Lacate-Plus meter (Nova Biomedical). The procedure is as follows: Researcher will don protective gloves prior to blood collection; using a finger of subject's choice, the finger will be thoroughly cleaned with an alcohol pad and lanced; with a collection strip inserted into the meter, blood from the lancing will be collected and read by the meter; subject's finger will be cleaned with a sterile gauze and all biohazard material will be disposed of according to local, state and federal biohazard guidelines. 2 meters will be used to collect a duplicate reading. This will be collected before the bench press protocols and then again after.
Changes in Psychomotor Vigilance Test | Performed one time at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3), once at the beginning of the session and then again at the end of the session.
  This test measures how quickly and accurately you can respond to simple tasks, like pressing a button when you see a specific symbol. It assesses your reaction time and attention span. Participants are instructed to press the <Spacebar> as fast as possible after a red stopwatch appears on screen. A valid response (response occurs after a stopwatch appears) is followed by reaction time feedback.
Perceived Recovery Status (PRS) Likert Scale | Performed at the beginning of Visits 2 and 3 (days 28 and 29) and then as the only outcome for Visit 4 (day 30).
  The PRS is a composite scale directly proportional to recovery (Laurent, et al. 2011). Hence, the purpose of the scale will be to assess the participant's recovery from the previous exercise session. Subjects will be informed that having no soreness and a high feeling of recovery is a 10, while extreme soreness and low feelings of recovery, leading to limited ability to function, is defined by a range of 0-3, adequate recovery, with some ability to function, is defined by a range of 4-7, and good recovery, with the ability to function normally, is defined by a range of 8-10.
Upper Body Soreness Likert Scale | Performed at the beginning of Visits 2 and 3 (days 28 and 29) and then as the only outcome for Visit 4 (day 30).
  A 7-point likert scale will be used for upper body muscle soreness, after performing 5 bodyweight pushups (modified for women, standard for men). The likert scale is a validated instrument designed to assess self reported muscle soreness, measured across a 7-point scale. The scale ranges from 0 (no soreness), to 6 (unbearable soreness), and has good validity and reliability (Impellizzeri, F., et al., 2007).
Estimated VO2max | Performed one time at baseline (visit 1), at day 28 (visit 2), and day 29 (visit 3).
  The total time taken to complete the 1 mile will be recorded as the primary performance measure. VO2max will be calculated from previously validated equations (Kayihan et al., 2014). This will be calculated at baseline and used to compare to subsequent visit testing for changes in aerobic capacity.

OTHER OUTCOMES:
Adverse Events | Continuously throughout the trial, up to 7 months.
  Will be recorded based on observation and verbal subject questioning. Defined as participants self-reported adverse effects. Items that will be surveyed include, but not limited to, headache, dizziness, nausea, vomiting, indigestion, blurred vision, lethargy, swelling, itching, chest pain, heart palpitations, difficulty breathing, lethargy, and muscle pain/cramps.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sikorski, PhD, Principal Investigator — Applied Science and Performance Institute
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macarilla CT, Sautter NM, Robinson ZP, Juber MC, Hickmott LM, Cerminaro RM, Benitez B, Carzoli JP, Bazyler CD, Zoeller RF, Whitehurst M, Zourdos MC. Accuracy of Predicting One-Repetition Maximum from Submaximal Velocity in The Barbell Back Squat and Bench Press. J Hum Kinet. 2022 Apr 26;82:201-212. doi: 10.2478/hukin-2022-0046. eCollection 2022 Apr. PMID 36196346
- [Background] Kayihan G, Ozkan A, Koklu Y, Eyuboglu E, Akca F, Koz M, Ersoz G. Comparative analysis of the 1-mile run test evaluation formulae: assessment of aerobic capacity in male law enforcement officers aged 20-23 years. Int J Occup Med Environ Health. 2014 Apr;27(2):165-74. doi: 10.2478/s13382-014-0237-0. Epub 2014 Feb 12. PMID 24519369
- [Background] Bradshaw DI, George JD, Hyde A, LaMonte MJ, Vehrs PR, Hager RL, Yanowitz FG. An accurate VO2max nonexercise regression model for 18-65-year-old adults. Res Q Exerc Sport. 2005 Dec;76(4):426-32. doi: 10.1080/02701367.2005.10599315. PMID 16739680
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893